CLINICAL TRIAL: NCT05332990
Title: Multicenter Comparison of Interictal High Frequency Oscillations as a Predictor of Seizure Freedom
Brief Title: Multicenter Comparison of Interictal HFO as a Predictor of Seizure Freedom
Acronym: multiHFO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Collaborators: McGill University (Other); University of Michigan (Other); University of Calgary (Other); Cook Children's Health Care System (Other); St. Anne's University Hospital Brno, Czech Republic (Other); Mayo Clinic (Other); Thomas Jefferson University (Other); UMC Utrecht (Other); Schweizerisches Epilepsie Zentrum (Unknown)
Responsible Party: Sponsor
Other Study IDs: multiHFO
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HFO analysis — We use an automated data-independent prospective definition of clinically relevant HFO that has been validated in data from two independent epilepsy centers.

SUMMARY:
In drug-resistant focal epilepsy, interictal high frequency oscillations (HFO) recorded from intracranial EEG (iEEG) may provide clinical information for delineating epileptogenic brain tissue. The iEEG electrode contacts that contain HFO are hypothesized to delineate the epileptogenic zone; their resection should then lead to postsurgical seizure freedom.

We test whether our prospective definition of clinically relevant HFO is in agreement with postsurgical seizure outcome. The algorithm is fully automated and is equally applied to all datasets. The aim is to assess the reliability of the proposed detector and analysis approach.

DETAILED DESCRIPTION:
We use an automated data-independent prospective definition of clinically relevant HFO that has been validated in data from two independent epilepsy centers. In this study, we combine retrospectively collected datasets from 9 independent epilepsy centers. The analysis is blinded to clinical outcome. We use iEEG recordings during NREM sleep with a minimum of 12 epochs of 5 minutes of NREM sleep. We automatically detect HFO in the ripple (80-250 Hz) and in the fast ripple (250-500 Hz) band. There is no manual rejection of events in this fully automated algorithm. The type of HFO that we consider clinically relevant is defined as the simultaneous occurrence of a fast-ripple and a ripple. We calculate the temporal consistency of each patient's HFO rates over several data epochs within and between nights. Patients with temporal consistency < 50% are excluded from further analysis. We determine whether all electrode contacts with high HFO rate are included in the resection volume and whether seizure freedom (ILAE 1) was achieved at ≥2 y follow-up.

Applying a previously validated algorithm to a large cohort from several independent epilepsy centers may advance the clinical relevance and the generalizability of HFO analysis as essential next step for use of HFO in clinical practice.

ELIGIBILITY:
Data as provided from the participating center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We include patients with drug-resistant focal epilepsy of all ages who 1) underwent invasive EEG recordings with subdural and/or depth electrodes as part of their pre-surgical evaluation 4, 2) underwent epilepsy surgery aiming at seizure freedom after resection of a single focus, and 3) and the postsurgical seizure outcome was determined by follow-up visits at ≥ 2 y 32. According to the International League Against Epilepsy (ILAE) Classification 3 we classify outcome into seizure freedom (ILAE 1) or recurrent seizures (ILAE 2-6). Outcome data that are assessed with the Engel scale are mapped to ILAE 1 or ILAE 2-6 respectively.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
seizure freedom | 2 years after surgery
  ILAE grade 1
seizure recurrence | within 2 years after surgery
  ILAE grade 2-6

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Neurosurgery, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dimakopoulos V, Gotman J, Stacey W, von Ellenrieder N, Jacobs J, Papadelis C, Cimbalnik J, Worrell G, Sperling MR, Zijlmans M, Imbach L, Frauscher B, Sarnthein J. Protocol for multicentre comparison of interictal high-frequency oscillations as a predictor of seizure freedom. Brain Commun. 2022 Jun 9;4(3):fcac151. doi: 10.1093/braincomms/fcac151. eCollection 2022. PMID 35770134
- [Result] Dimakopoulos V, Megevand P, Boran E, Momjian S, Seeck M, Vulliemoz S, Sarnthein J. Blinded study: prospectively defined high-frequency oscillations predict seizure outcome in individual patients. Brain Commun. 2021 Sep 2;3(3):fcab209. doi: 10.1093/braincomms/fcab209. eCollection 2021. PMID 34541534
- [Result] Fedele T, Burnos S, Boran E, Krayenbuhl N, Hilfiker P, Grunwald T, Sarnthein J. Resection of high frequency oscillations predicts seizure outcome in the individual patient. Sci Rep. 2017 Oct 23;7(1):13836. doi: 10.1038/s41598-017-13064-1. PMID 29062105
- [Derived] Dimakopoulos V, Gotman J, Klimes P, von Ellenrieder N, Tan SB, Smith G, Gliske SV, Maltseva M, Manalo MK, Pail M, Brazdil M, van Blooijs D, van 't Klooster MA, Johnson S, Laboy S, Ledergerber D, Imbach L, Papadelis C, Sperling MR, Zijlmans M, Cimbalnik J, Jacobs J, Stacey WC, Frauscher B, Sarnthein J. Multicentre analysis of seizure outcome predicted by removal of high-frequency oscillations. Brain. 2025 May 13;148(5):1769-1777. doi: 10.1093/brain/awae361. PMID 39530262
- See also: HFO analysis: publications, algorithms and data — https://hfozuri.ch/